CLINICAL TRIAL: NCT05555914
Title: Functional Evaluation of the Recovery of Prehension in Persons With Tetraplegia by Implanted Neural Stimulation
Brief Title: Neural Stimulation for Hand Grasp in People With Tetraplegia
Acronym: AGILIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Bouffard Vercelli - USSAP (Other)
Collaborators: Institut National de Recherche en Informatique et en Automatique (Other); NEURINNOV (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-A00205-38
Record Dates: First submitted 2022-08-29; First posted 2022-09-27 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2022-10

CONDITIONS: Tetraplegia
Keywords: Tetraplegia; Neural stimulation
MeSH Terms: conditions — Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurostimulation (Experimental): Implantation of 3 multicontact cuff electrodes in the upper limb of patients with tetraplegia
  Interventions: Other: Neurostimulation

INTERVENTIONS:
Other: Neurostimulation — Implantation of 3 multicontact cuff electrodes in the upper limb of patients with tetraplegia and control of the stimulation by contralateral shoulder movements

SUMMARY:
A selective neural stimulation as the investigators propose allows to stimulate several muscles via a single electrode. Neural stimulation requires less energy for muscle activation. In our approach, 2 electrodes will be implanted above the elbow on the median, the ulnar and the radial nerves. This considerably reduces the number of implanted elements and therefore i) the risk of infection, ii) the risk of failure, iii) the surgical risk through minimally invasive surgery.

Our main hypothesis is that multipolar neural electrical stimulation of the median and the ulnar nerve (flexion) and the radial nerve (extension) allows:

* on the one hand, a selective, individualized motor activation (muscle by muscle)
* on the other hand, a synergistic motor activation (association of several muscles) for the purpose of production of functional movements.

DETAILED DESCRIPTION:
Electrical stimulation of the muscles has been used for decades in rehabilitation units specializing in the treatment of spinal cord injuries. It has been shown to be effective in building muscle and preventing muscle atrophy following spinal cord injury (SCI) or stroke. It can also be used to reduce spasticity and above all to promote functionally useful motor control. It is then a Functional Electric Stimulation (FES). In the quadriplegic person marked by a severe motor deficiency of the upper limbs, FES is today the only technique allowing to restore a functional gripping movements in the case where the active muscular resources below the elbows are missing or too weak to allow tendon transfer surgery.

Like "Freehand", all the devices using FES directly stimulate the muscles (surface, intramuscular or epimysial electrodes) and therefore require a high number of internal components with a theoretical risk of infection and greater rejection. since each muscle must be activated via an electrode (up to 12 in the case of "FreeHand"). The investigators propose instead selective neural stimulation as it allows stimulating several muscles via a single electrode. Neural stimulation requires less energy for muscle activation. In our approach, three electrodes will be implanted above the elbow on the median, the ulnar and the radial nerves. This considerably reduces the number of implanted elements and therefore i) the risk of infection, ii) the risk of failure, iii) the surgical risk thanks to minimally invasive surgery. The procedure consisted of placing a multi-contact cuff electrode around the radial, ulnar or median nerves and observing the effects of electrical neural stimulation in terms of muscle selectivity, force produced and movement induced. In a previous study, the investigators already proved through acute intra operative testing (under Ethics Committee approval, #NCT03721861) that:

No failure of the electrodes or of the stimulator was noted. For all of the 8 subjects, it was possible to selectively stimulate muscle groups to obtain the opening of the thumb and fingers, or the flexion of the thumb, fingers and obtaining possibly functional grip like the forceps with opposition of the thumb or palmar grip.

A second feasibility study (Ethics committee registration #2016-A00711-50) with 17 quadriplegic patients assessed the subject's ability to use voluntary contractions of sus lesional muscles (EMG recordings in 8 subjects) or voluntary movements of shoulders (inertial recordings in 9 subjects) to control the movements of a robotic hand or the triggering of an electrical surface stimulation of the muscles of the forearm. All of the patients managed to master the proposed interface after a short familiarization period.

On the basis of the results of these two studies, the investigator wish to take an additional step in the development of a gripping assistance device for patients with spinal cord injury by proposing the implantation of three cuff electrodes with percutaneous connection on the arm of people with tetraplegia. The electrodes will be kept in place for a period of 1 month before being definitively explanted. An implanted cable will connect the electrodes to an external connector. A preliminary study based on the implantation of only 2 electrodes (on the median and the radial nerve) was conducted in 2020 in 2 patients.vNeither of the 2 participants showed general and local comorbidity. Acceptability was optimal. None of the stimulation configurations generated contradictory movements. The success rate in task execution by the electro-stimulated hand exceeded the target of 50% (54% and 51% for patient 1 and 2 respectively). The compliance rate of the control orders in both patients was > 90% using motion IMU-based detection and 100% using EMG-based detection in patient 1. These results support the relevance of neural stimulation of the tetraplegic upper limb with a more selective approach, using multi-contact epineural electrodes with 9 and 6 contact points for the median and radial nerve respectively.

ELIGIBILITY:
Inclusion Criteria

1. Informed consent signed
2. Patient affiliated to a social security (state medical aid excepted).
3. Neurological level ≥ C7 4.18 years old ≤ age ≤ 65 years old,

5.complete traumatic injury: defined by an A or B score on the AIS scale. (AIS A or - complete motor deficit under injury. This is an internationally agreed standard for describing spinal cord injury) 6.neurological stability (no change in muscle testing) > 6 months, 7.post-injury duration > 6 months 8.patients without active muscle resources for conventional tendon transfer surgery on the forearm and hand

Exclusion Criteria:

1. patient deprived of liberty (by judicial or administrative decision).
2. adult patient who is subject to a legal protection measure or unable to express consent
3. participation in another ongoing clinical trial
4. pregnant or breastfeeding women or women of childbearing age without effective contraception
5. spasticity and contractures in flexion or extension of the upper limbs of a destabilizing nature.
6. unstable epilepsy with a notion of a epileptic seizure that occurred within the previous 12 months.
7. unstable cardiovascular pathology (coronary heart disease, major hypertension, heart failure, etc.).
8. infectious pathology under treatment at the inclusion visit
9. wearing a pacemaker or a spinal cord stimulator implant
10. dermatological problems contraindicating the application of surface electrodes.
11. body weight >100 kg
12. psychiatric condition and/or history contraindicating participation in research
13. any contraindications to anesthesia and/or surgery
14. hypersensitivity to low molecular weight heparin (LMWH) or to any of the excipients of the specialty used
15. history of immune-mediated heparin-induced thrombocytopenia (HIT) within the last 100 days or presence of circulating antibodies
16. clinically significant active bleeding or a condition associated with a high risk of bleeding
17. electrical mapping identified as negative during the inclusion visit, i.e. with muscles revealing a rating < 4 MRC for at least one of the extensors (ECRL, ECRB, EDC, EPL) or one of the flexors (FPL, FDS, FDP).
18. bone fracture on the upper limbs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Functional outcome: Number of successful trials (task completed) out of 5 trials with 5 preselected objects. | Baseline prior to surgery and following surgery: Day5, Day6, Day8, Day12, Day15, Day17, Day22, Day26 and Day29
  The objective is to show that neural electrical stimulation allows the user to master the completion of each of pre-selected gripping tasks.
  The evaluation criteria is the number of successful trials (task completed) out of 5 trials with 5 preselected objects. For each object, a successful gripping task is a task completed in a duration <180 sec.

SECONDARY OUTCOMES:
Functional outcome | Following surgery from Day12: Day12, Day15, Day17, Day22, Day26 and Day29
  Evaluation of the patient's ability to perform functional takes (gripping, moving, letting go) of 5 objects chosen by the user, by means of multi-contact neural stimulation of the median, ulnar and radial nerves.
  Evaluation criterion: Canadian Occupational Performance Measure (COPM)
Strength | Baseline prior to surgery and following surgery: Day5, Day6, Day8, Day12, Day15, Day17, Day22, Day26 and Day29
  Measurements at the beginning and end of each session, in order to follow the exhaustion of the force produced over the course of the tests.
  The grip force is measured for 5 seconds with two gauges for each of the 2 takes three times in a row before any evaluation of the gripping tasks and 3 times in a row at the end of the 5 objects X 5 gripping tests. The average of the 3 measures is retained Evaluation criterion: Grip strength test and pinch grip test (dynamometer)
Fatigue | Baseline prior to surgery and following surgery: Day5, Day6, Day8, Day12, Day15, Day17, Day22, Day26 and Day29
  To measure a person's perception of his efforts and exertion and fatigue during each trial.
  Evaluation criterion: Borg test
Self perception and psychological well being | Baseline prior to surgery and following surgery: Day8, Day15, Day22, Day29
  To measure a person's perception of his well being. Evaluation criterion: The 5-item World Health Organization Well-Being Index (WHO-5)
System Usability Scale | Following surgery : Day8 and Day29
  To measure the potential usability of FES and the satisfaction provided by the use of the implanted electrical stimulation Evaluation criterion: The System Usability Scale (SUS).
  SUS scores have a range of 0 to 100. Scores for individual items are not meaningful on their own.The higher the score, the higher the perceived usability.
Local tolerance | Following surgery: daily from Day0 to Day29
  From the skin point of view, to look for an allergic and / or infectious dermatological lesion at the implantation site. The answer provided daily will be binary yes / no.
Pain assessment using the Visual Analog Scale (VAS) | Baseline prior to surgery and following surgery: Day5, Day6, Day8, Day12, Day15, Day17, Day22, Day26 and Day29
  From an algological point of view, assessment of the emergence or worsening of pain (score above 3/10 on the Analog Pain Scale) or a mean score above 3/10.

CONTACTS AND LOCATIONS:
Overall Officials: Charles FATTAL, MD, PhD, Principal Investigator — Centre Bouffard Vercelli - USSAP
Locations (1):
- Rehabilitation Center Bouffard-Vercelli USSAP, Perpignan, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fattal C, Teissier J, Geffrier A, Fonseca L, William L, Andreu D, Guiraud D, Azevedo-Coste C. Restoring Hand Functions in People with Tetraplegia through Multi-Contact, Fascicular, and Auto-Pilot Stimulation: A Proof-of-Concept Demonstration. J Neurotrauma. 2022 May;39(9-10):627-638. doi: 10.1089/neu.2021.0381. Epub 2022 Feb 2. PMID 35029125